CLINICAL TRIAL: NCT02340312
Title: Evaluation of the Duodenal Microbiome in Pediatric Functional Dyspepsia
Brief Title: Functional Dyspepsia Microbiome Study
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Craig A. Friesen, MD, M.D. Divison Cheif Gastroenterology, Children's Mercy Hospital Kansas City
Other Study IDs: 490390
Record Dates: First submitted 2014-12-15; First posted 2015-01-16 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Functional Dyspepsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collection of .5 aggregate of doudenal tissue. Collection of stool samples.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: EGD — In this study patients are being scoped(EGD) as standard of care and being asked to allow .5 aggregate of tissue biopsy to be taken for research purposes.
Other: Collection of Stool Specimens — We will be collecting stool samples from each participant for research purposes. Within two weeks after EGD tissue collection.

SUMMARY:
Recurrent abdominal pain has long been acknowledged to be the most common chronic pain entities in children. The purpose of this study is to describe the microbiome in children with FD and to explore relationships between the microbiome and postprandial distress syndrome, anxiety scores, and mucosal biomarkers or anxiety. The specific goals of this study are to: 1) Determine the frequencies and relative proportions for specific bacteria or bacteria phyla in children with FD in both duodenal mucosal specimens and stool samples. 2) Determine if the frequencies or proportions of specific bacteria or bacteria phyla differ between children with and without PDS. 3) Determine bi-variate correlations between bacteria/phyla frequency, bacteria/phyla proportions, anxiety scores, and mucosal biomarkers, respectively.

DETAILED DESCRIPTION:
The purpose of the current study is to describe the microbiome in children with FD and to explore relationships between the microbiome and postprandial distress syndrome, anxiety scores, and mucosal biomarkers or anxiety.

SPECIFIC AIMS

1. To determine the frequencies and relative proportions for specific bacteria or bacteria phyla in children with FD in both duodenal mucosal specimens and stool samples.
2. To determine if the frequencies or proportions of specific bacteria or bacteria phyla differ between children with and without PDS.
3. To determine bi-variate correlations between bacteria/phyla frequency, bacteria/ phyla proportion, anxiety scores, and mucosal biomarkers, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of FD as determined by the GI physician in accordance with Rome III criteria
* Age 8-17 years inclusive
* Scheduled for upper endoscopy as part of routine care after failing to respond to acid suppression therapy

Exclusion Criteria:

* Use of oral antibiotic or probiotic within 8 weeks prior to enrollment
* Use of systemic steroid or immunomodulating drug within 8 weeks of enrollment

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and adolecents ages 8 to 17 inclusive that have been diagonsed with functional dyspepsia and are scheduled to have a EGD with biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-01; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Microbiome Analysis | within 12 months from collection
  Fecal samples and 8 mucosal biopsies (descending duodenum) will be obtained from each subject. Samples will be processed and DNA isolated per standard lab techniques.16S rDNA sequence analysis of microbial communities within patient samples will be analyzed utilizing our HiSeq 1500 rapid run technologies. We will perform 2 X 150 bp paired end sequencing which will give exceptional coverage (reads > 30,000). We will sequence the V4 region of 16s RNA (E. coli 515-806), which is the method optimized for Illumina HiSeq 1500 currently. We will also sequence simultaneously the V3 region of 16s RNA to provide a dual-control analysis of samples. Confirmatory PCR will be employed when appropriate. Data will be reported as total counts for each identified bacterial species.
Inflammatory Cell Density | within 12 months from collection
  Routine histology slides previously stained with hematoxylin and eosin will be utilized for determination of eosinophil density.
  IHC techniques will be utilized for determination of mast cell density. Serial 3-μm paraffin sections will be air dried and heat fixed on slides. The sections will be deparaffinized with xylene and iodine and rehydrated in a graded series of alcohol. Utilizing tryptase monoclonal mouse antihuman mast cell tryptase antibody (clone AA1, Dako, Carpinteria, CA), sections will be stained on an automated Dako Autostainer 3400 using Dako's LSAB+ kit with streptavidin conjugated to horseradish peroxidase.
  To determine density for each cell type, the entire specimen will be scanned to determine the subjective area of greatest involvement. Density will be determined by counting cells within 5 consecutive high-power fields (400X magnification). Peak and mean cell densities expressed as cells/hpf will be determined. This will be completed before study end.
Immunohistochemistry (IHC) | within 12 months from collection
  IHC staining will be performed and may include DCLK1, BDNF, TRPV1, and/or CRH-R1, respectively, depending on the results of an on-going pilot study. Staining intensity will be evaluated in a blinded fashion by a pathologist to assign scores for average IHC signal intensity (i.e. 0= none, 1= mild, 2= moderate, and 3= strong) as well as the percentage of tissue cells or fibers showing positive immunoreactivity. A sem-quantitative scoring system will be applied in which the final immunoreactive score will equal the product of the percentage of positive cells times the average staining intensity. Percentage of positive cells or fibers will be graded as follows: 0= negative-10%, 1= 11-33%, 2= 33-66%, and 3= > 67%. Immunoreactivity will be considered positive when the combined score ranges between 2-6 and negative with a score of 0-1. Other IHC stains may be performed should they become relevant as indicated by the literature. This will be performed before study end.

SECONDARY OUTCOMES:
T-scores for the BASC will be collected as part of this study on the Data Collection Form. | within 6 months from completion
  This information is used to assess psychosocial information from the patient.This will be collected and recorded before study end.

CONTACTS AND LOCATIONS:
Overall Officials: Craig A Friesen, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- The Children's Mercy Hospital, Kansas City, Missouri, United States

REFERENCES:
- [Background] Hyams JS, Davis P, Sylvester FA, Zeiter DK, Justinich CJ, Lerer T. Dyspepsia in children and adolescents: a prospective study. J Pediatr Gastroenterol Nutr. 2000 Apr;30(4):413-8. doi: 10.1097/00005176-200004000-00012. PMID 10776953
- [Background] Youssef NN, Murphy TG, Langseder AL, Rosh JR. Quality of life for children with functional abdominal pain: a comparison study of patients' and parents' perceptions. Pediatrics. 2006 Jan;117(1):54-9. doi: 10.1542/peds.2005-0114. PMID 16396860
- [Background] Walker LS, Garber J, Van Slyke DA, Greene JW. Long-term health outcomes in patients with recurrent abdominal pain. J Pediatr Psychol. 1995 Apr;20(2):233-45. doi: 10.1093/jpepsy/20.2.233. PMID 7760222
- [Background] Gieteling MJ, Bierma-Zeinstra SM, Passchier J, Berger MY. Prognosis of chronic or recurrent abdominal pain in children. J Pediatr Gastroenterol Nutr. 2008 Sep;47(3):316-26. doi: 10.1097/MPG.0b013e31815bc1c1. PMID 18728528
- [Background] Schurman JV, Friesen CA, Danda CE, Andre L, Welchert E, Lavenbarg T, Cocjin JT, Hyman PE. Diagnosing functional abdominal pain with the Rome II criteria: parent, child, and clinician agreement. J Pediatr Gastroenterol Nutr. 2005 Sep;41(3):291-5. doi: 10.1097/01.mpg.0000178438.64675.c4. PMID 16131983
- [Background] Rasquin A, Di Lorenzo C, Forbes D, Guiraldes E, Hyams JS, Staiano A, Walker LS. Childhood functional gastrointestinal disorders: child/adolescent. Gastroenterology. 2006 Apr;130(5):1527-37. doi: 10.1053/j.gastro.2005.08.063. PMID 16678566
- [Background] Schurman JV, Singh M, Singh V, Neilan N, Friesen CA. Symptoms and subtypes in pediatric functional dyspepsia: relation to mucosal inflammation and psychological functioning. J Pediatr Gastroenterol Nutr. 2010 Sep;51(3):298-303. doi: 10.1097/MPG.0b013e3181d1363c. PMID 20479684
- [Background] Grenham S, Clarke G, Cryan JF, Dinan TG. Brain-gut-microbe communication in health and disease. Front Physiol. 2011 Dec 7;2:94. doi: 10.3389/fphys.2011.00094. eCollection 2011. PMID 22162969
- [Background] Konturek PC, Brzozowski T, Konturek SJ. Stress and the gut: pathophysiology, clinical consequences, diagnostic approach and treatment options. J Physiol Pharmacol. 2011 Dec;62(6):591-9. PMID 22314561
- [Background] Neufeld KM, Kang N, Bienenstock J, Foster JA. Reduced anxiety-like behavior and central neurochemical change in germ-free mice. Neurogastroenterol Motil. 2011 Mar;23(3):255-64, e119. doi: 10.1111/j.1365-2982.2010.01620.x. Epub 2010 Nov 5. PMID 21054680
- [Background] Rao AV, Bested AC, Beaulne TM, Katzman MA, Iorio C, Berardi JM, Logan AC. A randomized, double-blind, placebo-controlled pilot study of a probiotic in emotional symptoms of chronic fatigue syndrome. Gut Pathog. 2009 Mar 19;1(1):6. doi: 10.1186/1757-4749-1-6. PMID 19338686
- [Background] Cryan JF, O'Mahony SM. The microbiome-gut-brain axis: from bowel to behavior. Neurogastroenterol Motil. 2011 Mar;23(3):187-92. doi: 10.1111/j.1365-2982.2010.01664.x. PMID 21303428
- [Background] Lyte M, Li W, Opitz N, Gaykema RP, Goehler LE. Induction of anxiety-like behavior in mice during the initial stages of infection with the agent of murine colonic hyperplasia Citrobacter rodentium. Physiol Behav. 2006 Oct 30;89(3):350-7. doi: 10.1016/j.physbeh.2006.06.019. Epub 2006 Aug 2. PMID 16887154
- [Background] Gabel LA, Marin I, LoTurco JJ, Che A, Murphy C, Manglani M, Kass S. Mutation of the dyslexia-associated gene Dcdc2 impairs LTM and visuo-spatial performance in mice. Genes Brain Behav. 2011 Nov;10(8):868-75. doi: 10.1111/j.1601-183X.2011.00727.x. Epub 2011 Oct 19. PMID 21883923
- [Background] Li Y, Ji YJ, Jiang H, Liu DX, Zhang Q, Fan SJ, Pan F. Effects of unpredictable chronic stress on behavior and brain-derived neurotrophic factor expression in CA3 subfield and dentate gyrus of the hippocampus in different aged rats. Chin Med J (Engl). 2009 Jul 5;122(13):1564-9. PMID 19719949
- [Background] Shi SS, Shao SH, Yuan BP, Pan F, Li ZL. Acute stress and chronic stress change brain-derived neurotrophic factor (BDNF) and tyrosine kinase-coupled receptor (TrkB) expression in both young and aged rat hippocampus. Yonsei Med J. 2010 Sep;51(5):661-71. doi: 10.3349/ymj.2010.51.5.661. PMID 20635439
- [Background] Yang J, Yu Y, Yu H, Zuo X, Liu C, Gao L, Chen ZY, Li Y. The role of brain-derived neurotrophic factor in experimental inflammation of mouse gut. Eur J Pain. 2010 Jul;14(6):574-9. doi: 10.1016/j.ejpain.2009.10.007. Epub 2009 Nov 20. PMID 19932037
- [Background] Yu YB, Zuo XL, Zhao QJ, Chen FX, Yang J, Dong YY, Wang P, Li YQ. Brain-derived neurotrophic factor contributes to abdominal pain in irritable bowel syndrome. Gut. 2012 May;61(5):685-94. doi: 10.1136/gutjnl-2011-300265. Epub 2011 Oct 13. PMID 21997550
- [Background] Akbar A, Yiangou Y, Facer P, Walters JR, Anand P, Ghosh S. Increased capsaicin receptor TRPV1-expressing sensory fibres in irritable bowel syndrome and their correlation with abdominal pain. Gut. 2008 Jul;57(7):923-9. doi: 10.1136/gut.2007.138982. Epub 2008 Feb 5. PMID 18252749
- [Background] Miranda A, Nordstrom E, Mannem A, Smith C, Banerjee B, Sengupta JN. The role of transient receptor potential vanilloid 1 in mechanical and chemical visceral hyperalgesia following experimental colitis. Neuroscience. 2007 Sep 21;148(4):1021-32. doi: 10.1016/j.neuroscience.2007.05.034. Epub 2007 Aug 23. PMID 17719181
- [Background] Matsumoto K, Lo MW, Hosoya T, Tashima K, Takayama H, Murayama T, Horie S. Experimental colitis alters expression of 5-HT receptors and transient receptor potential vanilloid 1 leading to visceral hypersensitivity in mice. Lab Invest. 2012 May;92(5):769-82. doi: 10.1038/labinvest.2012.14. Epub 2012 Feb 13. PMID 22330338
- [Background] Yang CQ, Wei YY, Zhong CJ, Duan LP. Essential role of mast cells in the visceral hyperalgesia induced by T. spiralis infection and stress in rats. Mediators Inflamm. 2012;2012:294070. doi: 10.1155/2012/294070. Epub 2012 Mar 7. PMID 22529522
- [Background] Akbar A, Yiangou Y, Facer P, Brydon WG, Walters JR, Anand P, Ghosh S. Expression of the TRPV1 receptor differs in quiescent inflammatory bowel disease with or without abdominal pain. Gut. 2010 Jun;59(6):767-74. doi: 10.1136/gut.2009.194449. PMID 20551462
- [Background] Fukudo S, Nomura T, Hongo M. Impact of corticotropin-releasing hormone on gastrointestinal motility and adrenocorticotropic hormone in normal controls and patients with irritable bowel syndrome. Gut. 1998 Jun;42(6):845-9. doi: 10.1136/gut.42.6.845. PMID 9691924
- [Background] Dinan TG, Quigley EM, Ahmed SM, Scully P, O'Brien S, O'Mahony L, O'Mahony S, Shanahan F, Keeling PW. Hypothalamic-pituitary-gut axis dysregulation in irritable bowel syndrome: plasma cytokines as a potential biomarker? Gastroenterology. 2006 Feb;130(2):304-11. doi: 10.1053/j.gastro.2005.11.033. PMID 16472586
- [Background] Posserud I, Agerforz P, Ekman R, Bjornsson ES, Abrahamsson H, Simren M. Altered visceral perceptual and neuroendocrine response in patients with irritable bowel syndrome during mental stress. Gut. 2004 Aug;53(8):1102-8. doi: 10.1136/gut.2003.017962. PMID 15247175
- [Background] Bohmelt AH, Nater UM, Franke S, Hellhammer DH, Ehlert U. Basal and stimulated hypothalamic-pituitary-adrenal axis activity in patients with functional gastrointestinal disorders and healthy controls. Psychosom Med. 2005 Mar-Apr;67(2):288-94. doi: 10.1097/01.psy.0000157064.72831.ba. PMID 15784796
- [Background] Dickhaus B, Mayer EA, Firooz N, Stains J, Conde F, Olivas TI, Fass R, Chang L, Mayer M, Naliboff BD. Irritable bowel syndrome patients show enhanced modulation of visceral perception by auditory stress. Am J Gastroenterol. 2003 Jan;98(1):135-43. doi: 10.1111/j.1572-0241.2003.07156.x. PMID 12526949
- [Background] La JH, Sung TS, Kim HJ, Kim TW, Kang TM, Yang IS. Peripheral corticotropin releasing hormone mediates post-inflammatory visceral hypersensitivity in rats. World J Gastroenterol. 2008 Feb 7;14(5):731-6. doi: 10.3748/wjg.14.731. PMID 18205263
- [Background] Wood JD. Enteric neuroimmunophysiology and pathophysiology. Gastroenterology. 2004 Aug;127(2):635-57. doi: 10.1053/j.gastro.2004.02.017. PMID 15300595
- [Background] He SH. Key role of mast cells and their major secretory products in inflammatory bowel disease. World J Gastroenterol. 2004 Feb 1;10(3):309-18. doi: 10.3748/wjg.v10.i3.309. PMID 14760748
- [Background] Hall W, Buckley M, Crotty P, O'Morain CA. Gastric mucosal mast cells are increased in Helicobacter pylori-negative functional dyspepsia. Clin Gastroenterol Hepatol. 2003 Sep;1(5):363-9. doi: 10.1053/s1542-3565(03)00184-8. PMID 15017654
- [Background] Friesen CA, Lin Z, Singh M, Singh V, Schurman JV, Burchell N, Cocjin JT, McCallum RW. Antral inflammatory cells, gastric emptying, and electrogastrography in pediatric functional dyspepsia. Dig Dis Sci. 2008 Oct;53(10):2634-40. doi: 10.1007/s10620-008-0207-0. Epub 2008 Mar 5. PMID 18320315
- [Background] Friesen CA, Lin Z, Hyman PE, Andre L, Welchert E, Schurman JV, Cocjin JT, Burchell N, Pulliam S, Moore A, Lavenbarg T, McCallum RW. Electrogastrography in pediatric functional dyspepsia: relationship to gastric emptying and symptom severity. J Pediatr Gastroenterol Nutr. 2006 Mar;42(3):265-9. doi: 10.1097/01.mpg.0000189367.99416.5e. PMID 16540794
- [Background] Santos J, Saperas E, Nogueiras C, Mourelle M, Antolin M, Cadahia A, Malagelada JR. Release of mast cell mediators into the jejunum by cold pain stress in humans. Gastroenterology. 1998 Apr;114(4):640-8. doi: 10.1016/s0016-5085(98)70577-3. PMID 9516384
- [Background] Friesen CA, Sandridge L, Andre L, Roberts CC, Abdel-Rahman SM. Mucosal eosinophilia and response to H1/H2 antagonist and cromolyn therapy in pediatric dyspepsia. Clin Pediatr (Phila). 2006 Mar;45(2):143-7. doi: 10.1177/000992280604500205. PMID 16528434
- [Background] Talley NJ, Walker MM, Aro P, Ronkainen J, Storskrubb T, Hindley LA, Harmsen WS, Zinsmeister AR, Agreus L. Non-ulcer dyspepsia and duodenal eosinophilia: an adult endoscopic population-based case-control study. Clin Gastroenterol Hepatol. 2007 Oct;5(10):1175-83. doi: 10.1016/j.cgh.2007.05.015. Epub 2007 Aug 7. PMID 17686660
- [Background] Friesen CA, Andre L, Garola R, Hodge C, Roberts C. Activated duodenal mucosal eosinophils in children with dyspepsia: a pilot transmission electron microscopic study. J Pediatr Gastroenterol Nutr. 2002 Sep;35(3):329-33. doi: 10.1097/00005176-200209000-00017. PMID 12352522
- [Background] Friesen CA, Kearns GL, Andre L, Neustrom M, Roberts CC, Abdel-Rahman SM. Clinical efficacy and pharmacokinetics of montelukast in dyspeptic children with duodenal eosinophilia. J Pediatr Gastroenterol Nutr. 2004 Mar;38(3):343-51. doi: 10.1097/00005176-200403000-00021. PMID 15076638
- [Background] Chrousos GP. Stress, chronic inflammation, and emotional and physical well-being: concurrent effects and chronic sequelae. J Allergy Clin Immunol. 2000 Nov;106(5 Suppl):S275-91. doi: 10.1067/mai.2000.110163. PMID 11080744
- [Background] Kokkotou E, Torres D, Moss AC, O'Brien M, Grigoriadis DE, Karalis K, Pothoulakis C. Corticotropin-releasing hormone receptor 2-deficient mice have reduced intestinal inflammatory responses. J Immunol. 2006 Sep 1;177(5):3355-61. doi: 10.4049/jimmunol.177.5.3355. PMID 16920976
- [Background] Leung L, Cahill CM. TNF-alpha and neuropathic pain--a review. J Neuroinflammation. 2010 Apr 16;7:27. doi: 10.1186/1742-2094-7-27. PMID 20398373
- [Background] White FA, Feldman P, Miller RJ. Chemokine signaling and the management of neuropathic pain. Mol Interv. 2009 Aug;9(4):188-95. doi: 10.1124/mi.9.4.7. PMID 19720751
- [Background] Edgar RC. Search and clustering orders of magnitude faster than BLAST. Bioinformatics. 2010 Oct 1;26(19):2460-1. doi: 10.1093/bioinformatics/btq461. Epub 2010 Aug 12. PMID 20709691
- [Background] DeSantis TZ, Hugenholtz P, Larsen N, Rojas M, Brodie EL, Keller K, Huber T, Dalevi D, Hu P, Andersen GL. Greengenes, a chimera-checked 16S rRNA gene database and workbench compatible with ARB. Appl Environ Microbiol. 2006 Jul;72(7):5069-72. doi: 10.1128/AEM.03006-05. PMID 16820507
- [Background] Caporaso JG, Bittinger K, Bushman FD, DeSantis TZ, Andersen GL, Knight R. PyNAST: a flexible tool for aligning sequences to a template alignment. Bioinformatics. 2010 Jan 15;26(2):266-7. doi: 10.1093/bioinformatics/btp636. Epub 2009 Nov 13. PMID 19914921
- [Background] Price MN, Dehal PS, Arkin AP. FastTree: computing large minimum evolution trees with profiles instead of a distance matrix. Mol Biol Evol. 2009 Jul;26(7):1641-50. doi: 10.1093/molbev/msp077. Epub 2009 Apr 17. PMID 19377059
- [Background] Helmus MR, Bland TJ, Williams CK, Ives AR. Phylogenetic measures of biodiversity. Am Nat. 2007 Mar;169(3):E68-83. doi: 10.1086/511334. Epub 2007 Jan 17. PMID 17230400
- [Background] Lozupone C, Lladser ME, Knights D, Stombaugh J, Knight R. UniFrac: an effective distance metric for microbial community comparison. ISME J. 2011 Feb;5(2):169-72. doi: 10.1038/ismej.2010.133. Epub 2010 Sep 9. No abstract available. PMID 20827291
- [Background] Lozupone C, Knight R. UniFrac: a new phylogenetic method for comparing microbial communities. Appl Environ Microbiol. 2005 Dec;71(12):8228-35. doi: 10.1128/AEM.71.12.8228-8235.2005. PMID 16332807
- [Background] Friesen CA, Schurman JV, Qadeer A, Andre L, Welchert E, Cocjin J. Relationship between mucosal eosinophils and anxiety in pediatric dyspepsia. Gastroenterology 2005; 129:A-158
- [Background] Carpenter S. That gut feeling. Monitor on Psychol 2012; 43:51-55
- [Background] Bienenstock J, Collins S. 99th Dahlem conference on infection, inflammation and chronic inflammatory disorders: psycho-neuroimmunology and the intestinal microbiota: clinical observations and basic mechanisms. Clin Exp Immunol. 2010 Apr;160(1):85-91. doi: 10.1111/j.1365-2249.2010.04124.x. PMID 20415856